CLINICAL TRIAL: NCT04554251
Title: Global Impact of COVID-19 on Pulmonology Special Units (Bronchoscopy, Thoracoscopy, Ultrasonography and Sleep Lab)
Brief Title: Global Impact of COVID-19 on Pulmonology Special Units
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aliae AR Mohamed Hussein, Professor of Pulmonology, Assiut University
Other Study IDs: Assiut20
Record Dates: First submitted 2020-09-06; First posted 2020-09-18 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Covid19; Global Impact; Pulmonology
Keywords: Bronchoscopy; Thoracoscopy; Thoracic ultrasonography; Sleep Lab; Global impact
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — invited questionnaire

SUMMARY:
The COVID-19 pandemic is having a profound impact on the world. As of May 18, 2020, there were 4,889,287 confirmed cases and 322,683 deaths globally. The healthcare system is wrestling with a virus that threatens to overwhelm hospital capacity, while simultaneously confronting an unprecedented reduction in elective and non-essential care.

A survey by the American Cancer Society showed that 50% of cancer patients and survivors reported some impact to their healthcare due to the COVID-19 epidemic.

A recent survey was conducted by Forbes et al to evaluate the changes in GI and endoscopy practices in North America.

However, the impact of this epidemic on Pulmonology units ( bronchoscopy, thoracoscopy, ultrsonography and sleep lab) globally has not been studied.

ELIGIBILITY:
Inclusion Criteria:

* Working registered invited pulmonology units; governmental, university, private

Exclusion Criteria:

* non pulmonary medicine registered units

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: invited pulmonology units; bronchoscopy, thoracoscopy, chest ultrasonography and sleep lab
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
global impact of COVID-19 on baseline patients number | 6 months
  number of patients and procedures before and after pandemic
measure the changes in practice in each unit | 6 months
  use of PPE
frequency of SARS-CoV-2 infection in healthcare workers | 6 months
  SARS-CoC-2 infection

CONTACTS AND LOCATIONS:
Overall Officials: Aliae Mohamed-Hussein, Study Chair — Assiut University
Locations (1):
- Aliae Mohamed-Hussein, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No